CLINICAL TRIAL: NCT00886340
Title: A Lifestyle Change Program to Prevent Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Robin Whittemore, Associate Professor, National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DK70594 (completed)
Record Dates: First submitted 2009-01-22; First posted 2009-04-22 (Estimated); Results first posted 2009-04-22 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-04

CONDITIONS: Prediabetes
Keywords: diabetes prevention, primary care
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced standard care (Active Comparator)
  Interventions: Behavioral: Enhanced standard care
- Lifestyle counseling (Experimental)
  Interventions: Behavioral: Lifestyle counseling

INTERVENTIONS:
Behavioral: Enhanced standard care — One appointment with nurse practitioner (20 minutes) One appointment with nutritionist (45 minutes)
  Arms: Enhanced standard care
Behavioral: Lifestyle counseling — Enhanced standard care Six appointments with nurse practitioner (20 minutes)
  Arms: Lifestyle counseling

SUMMARY:
The purpose of this study was to evaluate the effect of a diabetes prevention program provided by nurse practitioners in primary care to adults at risk for diabetes.

ELIGIBILITY:
Inclusion Criteria

* age 21 or older
* medically stable and safe to exercise
* at high risk for type 2 diabetes
* able to speak English.

Exclusion Criteria

* Type 2 diabetes
* Cardiovascular disease
* Cancer requiring treatment in the past 5 years
* Anemia
* Hepatitis
* Renal disease
* Gastrointestinal disease
* Recent or significant abdominal surgery
* Pulmonary disease with dependence on oxygen or daily use of bronchodilators
* Chronic infection (ie., HIV, active tuberculosis)
* Unable to walk 0.25 miles in 10 minutes
* Participation in commercial diet program
* Currently pregnant or within 3 months postpartum
* Currently nursing or within 6 weeks of having completed nursing
* Treatment of impaired glucose tolerance (IGT) with metformin
* Currently taking any glucocorticoid or beta-blocker
* Recently prescribed or changed dose of a statin (within 2 months)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2005-09; Primary Completion 2007-09 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin Whittemore, PhD, Principal Investigator — Yale School of Nursing

REFERENCES:
- [Result] Whittemore R, Melkus G, Wagner J, Dziura J, Northrup V, Grey M. Translating the diabetes prevention program to primary care: a pilot study. Nurs Res. 2009 Jan-Feb;58(1):2-12. doi: 10.1097/NNR.0b013e31818fcef3. PMID 19092550

RESULTS

PARTICIPANT FLOW:
Groups:
- Enhanced Standard Care: Enhanced standard care (one appointment with nurse practitioner and one appointment with nutritionist)
- Lifestyle Counseling: Lifestyle counseling (enhanced standard care and 6 appointments with nurse practitioner)
Period: Overall Study
Arm/Group | Enhanced Standard Care | Lifestyle Counseling
Started | 27 | 31
Completed | 27 | 24
Not Completed | 0 | 7
Not completed — Withdrawal by Subject | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Standard Care | Lifestyle Counseling | Total
Number analyzed (Participants) | 27 | 31 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 27 | 53
  >=65 years | 1 | 4 | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 43.2 (13.2) | 48.2 (12.4) | 45.7 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 28 | 52
  Male | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Met Weight Loss Goal of 5% Weight Loss
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Enhanced Standard Care | Lifestyle Counseling
Number analyzed (Participants) | 27 | 24
participants | 3 | 6
Statistical Analysis 1: Comparison: Enhanced Standard Care vs Lifestyle Counseling; pilot test, used 20% of sample required for a full test of the hypothesis; Test type: Superiority or Other; p = 0.08, Mixed Models Analysis — controlled for site, income, race/ethnicity

2. Secondary Outcome: Diet and Exercise Behavior
Time Frame: 6 months
Reporting Status: Not Posted

3. Secondary Outcome: Lipids
Time Frame: 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Quality of Life
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Enhanced Standard Care | Lifestyle Counseling
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/31
Other Adverse Events (participants affected / at risk) | 0/27 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No